CLINICAL TRIAL: NCT01120210
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Investigate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of JNJ-39588146 in Subjects With Heart Failure
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of an Intravenous Solution of JNJ-39588146 or Placebo in Patients With Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017116; 39588146AHF2001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); 2009-013929-42 (EudraCT Number); NCT01678768 (obsolete NCT alias)
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Results first posted 2013-06-25 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiac Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1 (Main Study) (Experimental): 3 consecutive 1-hour infusions of JNJ-39588146 5, 15, or 30 ng/kg/min or matching placebo
  Interventions: Drug: JNJ-39588146 5 ng/kg/min; Drug: JNJ-39588146 15 ng/kg/min; Drug: JNJ-39588146 30 ng/kg/min; Drug: Placebo
- Part 2 (Extended Infusion Sub-Study) (Experimental): 1 18-hr infusion of JNJ-39588146 of the highest tolerated dose from Part 1 of the study or matching placebo
  Interventions: Drug: Placebo; Drug: JNJ-39588146 5, 15, or 30 ng/kg/min

INTERVENTIONS:
Drug: JNJ-39588146 5 ng/kg/min — 1-hour infusion of JNJ-39588146 5 ng/kg/min on Day 1
  Arms: Part 1 (Main Study)
Drug: JNJ-39588146 15 ng/kg/min — 1-hour infusion of JNJ-39588146 15 ng/kg/min on Day 1
  Arms: Part 1 (Main Study)
Drug: JNJ-39588146 30 ng/kg/min — 1-hour infusion of JNJ-39588146 30 ng/kg/min on Day 1
  Arms: Part 1 (Main Study)
Drug: Placebo — 1-hour infusion of matching placebo on Day 1
Drug: JNJ-39588146 5, 15, or 30 ng/kg/min — 18-hour infusion of JNJ-39588146 or matching placebo on Day 1 immediately folllowing the 3-hour infusion at a dose equal to the maximum dose tolerated by that patient during the 3-hour infusion in Part 1 of the study.
  Arms: Part 2 (Extended Infusion Sub-Study)

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, pharmacodynamics (how the study medication affects the body) and pharmacokinetics (how the drug is absorbed in the body, how it is distributed within the body and removed from the body over time) of an intravenous administration of JNJ-39588146 or placebo over a 3-hour period in patients with heart failure. The highest tolerated dose received during the first 3 hours of the study will be administered to some patients for an additional 18 hours. There will be up to 3 doses given throughout the administration period over a total of up to 21 hours.

DETAILED DESCRIPTION:
This study will assess the safety, tolerability, pharmacodynamics and pharmacokinetics of JNJ-39588146 or placebo (which looks like the drug being studied but has no active ingredients) in patients with heart failure. This study is being conducted in two parts. Part 1 is a randomized (study drug will be assigned by chance), double-blind (neither the physician nor patient knows the identity of the assigned drug) study of 3 intravenous doses of JNJ-39588146 or placebo administered in 1-hr intervals (for a total of 3 hours) in 60 patients with heart failure. Part 2 is an extended infusion of JNJ-39588146 and placebo that will administer the highest tolerated dose from Part 1 for an additional 18 hours. The entire duration of the infusion could be as long as 21 hours. There is a 1 in 4 chance of getting placebo. The participation period is a maximum of 42 days, including a screening visit, a 2-day in-clinic period and two follow-up visits. For both parts of the study, patients will have a cardiac catheter in place to monitor heart function. Safety evaluations, which will include ECG (electrocardiograph, measuring the electrical currents in the heart), vital signs and monitoring of side-effects will be performed. Additionally, blood and urine samples will be collected for evaluation. Part 1: Patients will receive an intravenous (IV) solution of three different doses of JNJ-39588146 or placebo administered over 1 hour periods for a total of 3 hours. Part 2: Patients participating in the sub study will continue receiving an IV solution for 18 more hours for a total of up to 21 hours of administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with heart failure
* Women must be either postmenopausal or have been surgically sterilized at least 6 months ago
* Males must be willing to use an acceptable birth control method for 3 months after the last dose of study medication.

Exclusion Criteria:

* Patients must not have had an heart-assist device or heart transplant or be in imminent need of one
* Patients must not have had an ischemic attack within the last 6 months or a heart attack within the last month
* Patients must not have lung disease or congenital heart failure.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (9):
- Belgium (3):
  - Aalst
  - B-1070 Bruxelles
  - Genk
- Germany (2):
  - Bad Nauheim
  - Hamburg
- Poland (2):
  - Warsaw
  - Wroclaw
- Romania (2):
  - Bucharest
  - Tg. Mures

REFERENCES:
- [Derived] Gheorghiade M, Greene SJ, Ponikowski P, Maggioni AP, Korewicki J, Macarie C, Metra M, Grzybowski J, Bubenek-Turconi SI, Radziszewski W, Olson A, Bueno OF, Ghosh A, Deckelbaum LI, Li LY, Patel AR, Koester A, Konstam MA. Haemodynamic effects, safety, and pharmacokinetics of human stresscopin in heart failure with reduced ejection fraction. Eur J Heart Fail. 2013 Jun;15(6):679-89. doi: 10.1093/eurjhf/hft023. Epub 2013 Mar 6. PMID 23471413

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 5 countries: Belgium (3 sites), Germany (3 sites), Italy (5 sites), Poland (3 sites), and Romania (3 sites). A total of 62 subjects (16 subjects in the placebo group and 46 subjects in the JNJ-39588146 group) were randomized and treated with the study drug.
Pre-assignment Details: Patients had an option to participate in an 18 hour extended infusion sub-study following the initial 3-hour infusion main study with the highest dose. A total of 10 patients (7 patients in the JNJ-39588146 group and 3 patients in the placebo group) participated in the sub-study.
Groups:
- Placebo: Patients received 3 consecutive escalating intravenous (IV) infusions of placebo identical in appearance to JNJ-39588146. Each dose was planned to be infused over 1 hour for a total planned infusion time in the main study of 3 hours. Patients had an option to participate in an 18-hour extended infusion sub-study following the initial 3-hour infusion main study with the highest dose.
- JNJ-39588146: Patients received 3 consecutive escalating intravenous (IV) infusions of JNJ-39588146. Each dose was planned to be infused over 1 hour for a total planned infusion time in the main study of 3 hours. Patients had an option to participate in an 18-hour extended infusion sub-study following the initial 3-hour infusion main study with the highest dose.
Period: MAIN INFUSION
Arm/Group | Placebo | JNJ-39588146
Started | 16 | 46
Completed | 15 | 45
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: 18-HOUR EXTENDED INFUSION SUBSTUDY
Arm/Group | Placebo | JNJ-39588146
Started | 3 | 7
Completed | 3 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | JNJ-39588146 | Total
Number analyzed (Participants) | 16 | 46 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 35 | 46
  >=65 years | 5 | 11 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.46) | 56.6 (12.91) | 56.8 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 15 | 41 | 56
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 4 | 4
  Germany | 5 | 2 | 7
  Italy | 2 | 7 | 9
  Poland | 4 | 21 | 25
  Romania | 5 | 12 | 17
AgeCategorical [Number; unit: participants]
  <=10 years | 0 | 0 | 0
  11 - 20 years | 0 | 0 | 0
  21 - 50 years | 4 | 12 | 16
  50 - 64 years | 7 | 23 | 30
  >=65 years | 5 | 11 | 16

OUTCOME MEASURES:

1. Primary Outcome: Post-baseline Changes Compared to Placebo (at 1-, 2-, and 3-hours Post Infusion Initiation [ie, at the End of 5, 15 and 30 ng/kg/Min Infusions]) in Cardiac Index (CI)
Description: The effect of JNJ-39588146 on cardiac index (CI), a hemodynamic parameter that relates heart performance to the size of the individual measured in liters per minute per square metre (l/min/m2) was evaluated in patients with heart failure (HF). The primary analysis of this study focused on the differences between the treatment groups in terms of Least Squares (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from Baseline in CI at each time point as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: The modified intent-to-treat (MITT) population included all randomized patients who received at least 1 dose of study drug, had baseline measurement and at least 1 post-baseline measurement value of at least 1 of the primary endpoints. The efficacy analysis was to be performed using the MITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: L/min/m2
Groups:
- Placebo: Patients received 3 consecutive escalating intravenous (IV) infusions of placebo identical in appearance to JNJ-39588146. Each dose was planned to be infused over 1 hour for a total planned infusion time in the main study of 3 hours.
- JNJ-39588146: Patients received 3 consecutive escalating intravenous (IV) infusions of JNJ-39588146. Each dose was planned to be infused over 1 hour for a total planned infusion time in the main study of 3 hours. Planned doses were 5, 15 and 30 ng/kg/min.
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 16 | 46
L/min/m2
  1 hour infusion (5 ng/kg/min) | -0.03 (0.19) | 0.24 (0.14)
  2 hour infusion (15 ng/kg/min) | -0.15 (0.17) | 0.18 (0.13)
  3 hour infusion (30 ng/kg/min) | -0.05 (0.23) | 0.52 (0.17)
Statistical Analysis 1: Comparison: Placebo vs JNJ-39588146; 90% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in cardiac index (CI) at the end of the 5 ng/kg/min dose; Test type: Superiority or Other; p = 0.0595, ANCOVA; one-sided p-value and one-sided alpha=0.05; Mean Difference (Final Values) = 0.27, 90% CI 2-sided [-0.016 to 0.564]
Statistical Analysis 2: Comparison: Placebo vs JNJ-39588146; 90% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in cardiac index (CI) at the end of the 15 ng/kg/min dose; Test type: Superiority or Other; p = 0.0215, ANCOVA — one-sided p-value and one-sided alpha=0.05; Mean Difference (Final Values) = 0.33, 90% CI 2-sided [0.064 to 0.595]
Statistical Analysis 3: Comparison: Placebo vs JNJ-39588146; 90% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in cardiac index (CI) at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.0049, ANCOVA — one-sided p-value and one-sided alpha=0.05; Mean Difference (Final Values) = 0.57, 90% CI 2-sided [0.214 to 0.921]

2. Primary Outcome: Post-baseline Changes Compared to Placebo (at 1-, 2-, and 3-hours Post Infusion Initiation [ie, at the End of 5, 15 and 30 ng/kg/Min Infusions]) in Pulmonary Capillary Wedge Pressure (PCWP)
Description: The effect of JNJ-39588146 on pulmonary capillary wedge pressure (PCWP) was evaluated by administering multiple ascending doses of JNJ-39588146 or placebo over a 3-hour intravenous (IV) infusion period to patients with heart failure. The primary analysis of this study focused on the differences between the treatment groups in terms of Least Squares (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from baseline in PCWP at each time point as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 16 | 46
mmHg
  1 hour infusion (5 ng/kg/min) | -0.75 (1.43) [-2.312 to 2.131] | -0.84 (1.03)
  2 hour infusion (15 ng/kg/min) | 0.15 (1.81) [-4.164 to 1.464] | -1.20 (1.31)
  3 hour infusion (30 ng/kg/min) | 0.05 (1.97) [-5.639 to 0.483] | -2.53 (1.42)
Statistical Analysis 1: Comparison: Placebo vs JNJ-39588146; 90% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in pulmonary capillary wedge pressure (PCWP) at the end of the 5 ng/kg/min dose; Test type: Superiority or Other; p = 0.4729, ANCOVA — one-sided p-value and one-sided alpha=0.05; Mean Difference (Final Values) = -0.09, 90% CI 2-sided [-2.312 to 2.131]
Statistical Analysis 2: Comparison: Placebo vs JNJ-39588146; 90% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in pulmonary capillary wedge pressure (PCWP) at the end of the 15 ng/kg/min dose; Test type: Superiority or Other; p = 0.2123, ANCOVA — one-sided p-value and one-sided alpha=0.05; Mean Difference (Final Values) = -1.35, 90% CI 2-sided [-4.164 to 1.464]
Statistical Analysis 3: Comparison: Placebo vs JNJ-39588146; 90% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in pulmonary capillary wedge pressure (PCWP) at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.0821, ANCOVA — one-sided p-value and one-sided alpha=0.05; Mean Difference (Final Values) = -2.58, 90% CI 2-sided [-5.639 to 0.483]

3. Secondary Outcome: Post-baseline Changes Compared to Placebo (at 1-, 2-, and 3-hours Post Infusion Initiation [ie, at the End of 5, 15 and 30 ng/kg/Min Infusions]) in Heart Rate (HR)
Description: The primary analysis of this study focused on the differences between the treatment groups in terms of Least Squares (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from Baseline in heart rate (HR) at each time point as well as treatment group LS means and Standard Errors.
Time Frame: At 1-hour, 2 hours and 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 16 | 44
beats per minute (bpm)
  1 hour infusion (5 ng/kg/min) | 3.02 (1.24) [-2.527 to 1.879] | 2.69 (0.91)
  2 hour infusion (15 ng/kg/min) | 3.72 (1.69) [-1.764 to 4.235] | 4.96 (1.24)
  3 hour infusion (30 ng/kg/min) | 3.07 (1.81) [-1.046 to 5.372] | 5.23 (1.32)
Statistical Analysis 1: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in heart rate (HR) at the end of the 5 ng/kg/min dose; Test type: Superiority or Other; p = 0.7682, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-2.527 to 1.879]
Statistical Analysis 2: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in heart rate (HR) at the end of the 15 ng/kg/min dose; Test type: Superiority or Other; p = 0.4107, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = 1.24, 95% CI 2-sided [-1.764 to 4.235]
Statistical Analysis 3: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in heart rate (HR) at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.1811, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = 2.16, 95% CI 2-sided [-1.046 to 5.372]

4. Secondary Outcome: Post-baseline Changes Compared to Placebo (at 1-, 2-, and 3-hours Post Infusion Initiation [ie, at the End of 5, 15 and 30 ng/kg/Min Infusions]) in Systolic Blood Pressure (SBP)
Description: The primary analysis of this study focused on the differences between the treatment groups in terms of Least Squares (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from Baseline in systolic blood pressure (SBP) at each time point as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 16 | 46
mmHg
  1 hour infusion (5 ng/kg/min) | 0.15 (2.95) [-6.060 to 4.718] | -0.53 (2.12)
  2 hour infusion (15 ng/kg/min) | 6.94 (3.17) [-7.781 to 3.801] | 4.94 (2.28)
  3 hour infusion (30 ng/kg/min) | 6.32 (4.09) [-11.251 to 3.708] | 2.55 (2.94)
Statistical Analysis 1: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in systolic blood pressure (SBP) at the end of the 5 ng/kg/min dose; Test type: Superiority or Other; p = 0.8030, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-6.060 to 4.718]
Statistical Analysis 2: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in systolic blood pressure (SBP) at the end of the 15 ng/kg/min dose; Test type: Superiority or Other; p = 0.4923, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-7.781 to 3.801]
Statistical Analysis 3: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in systolic blood pressure (SBP) at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.3152, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -3.77, 95% CI 2-sided [-11.251 to 3.708]

5. Secondary Outcome: Post-baseline Changes Compared to Placebo (at 1-, 2-, and 3-hours Post Infusion Initiation [ie, at the End of 5, 15 and 30 ng/kg/Min Infusions]) in Diastolic Blood Pressure (DBP)
Description: The primary analysis of this study focused on the differences between the treatment groups in terms of LS mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in Least Square (LS) means (and associated confidence intervals) for change from Baseline in diastolic blood pressure(DBP) at each time point as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 16 | 46
mmHg
  1 hour infusion (5 ng/kg/min) | -0.43 (2.57) [-8.047 to 1.331] | -3.78 (1.83)
  2 hour infusion (15 ng/kg/min) | 1.83 (2.70) [-10.482 to -0.622] | -3.72 (1.93)
  3 hour infusion (30 ng/kg/min) | 3.05 (2.60) [-11.818 to -2.332] | -4.03 (1.86)
Statistical Analysis 1: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in diastolic blood pressure (DBP) at the end of the 5 ng/kg/min dose; Test type: Superiority or Other; p = 0.1561, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -3.36, 95% CI [-8.047 to 1.331]
Statistical Analysis 2: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in diastolic blood pressure (DBP) at the end of the 15 ng/kg/min dose; Test type: Superiority or Other; p = 0.0282, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -5.55, 95% CI 2-sided [-10.482 to -0.622]
Statistical Analysis 3: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in diastolic blood pressure (DBP) at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.0043, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -7.08, 95% CI 2-sided [-11.818 to -2.332]

6. Secondary Outcome: Post-baseline Changes Compared to Placebo (at 3-hours Post Infusion Initiation [ie, at the End of the 30 ng/kg/Min Infusion]) in Left Ventricular End Systolic Volume (LVESV)
Description: The primary analysis of this study focused on the differences between the treatment groups in terms of Least Squares (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from Baseline in left ventricular end systolic volume (LVESV) at the end of the 30 ng/kg/min infusion as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 12 | 36
mL | -15.51 (8.93) [-16.347 to 16.823] | -15.28 (6.36)
Statistical Analysis 1: Comparison: Placebo; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in left ventricular end systolic volume (LVESV) at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.9769, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-16.347 to 16.823]

7. Secondary Outcome: Post-baseline Changes Compared to Placebo (at 3-hours Post Infusion Initiation [ie, at the End of 30 ng/kg/Min Infusion]) in Left Ventricular End Diastolic Volume (LVEDV)
Description: The primary analysis of this study focused on the differences between the treatment groups in terms of Least Squares (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from Baseline in Left Ventricular End Diastolic Volume (LVEDV) at the end of the 30 ng/kg/min infusion as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 12 | 36
mL | -13.91 (10.05) [-16.592 to 20.551] | -11.93 (7.11)
Statistical Analysis 1: Comparison: Placebo; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in LVEDV at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.8297, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = 1.98, 95% CI 2-sided [-16.592 to 20.551]

8. Secondary Outcome: Post-baseline Changes Compared to Placebo (at 3-hours Post Infusion Initiation [ie, at the End of the 30 ng/kg/Min Infusion]) in Left Ventricular Ejection Fraction (LVEF)
Description: The primary analysis of this study focused on the differences between the treatment groups in terms of Least Squares (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from Baseline in Left Ventricular Ejection Fraction (LVEF) at the end of the 30 ng/kg/min infusion as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 12 | 36
percentage | 3.61 (1.93) [-3.352 to 3.968] | 3.92 (1.38)
Statistical Analysis 1: Comparison: Placebo; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in LVEF at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.8650, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-3.352 to 3.968]

9. Secondary Outcome: Post-baseline Changes Compared to Placebo (at 3-hours Post Infusion Initiation [ie, at the End of the 30 ng/kg/Min Infusion]) in Fractional Shortening (FS)
Description: The primary analysis of this study focused on the differences between the treatment groups in terms of Least Squares (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from Baseline in Fractional Shortening (FS) at the end of the 30 ng/kg/min infusion as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 13 | 33
percentage | 0.22 (1.54) [-1.204 to 3.102] | 1.17 (1.14)
Statistical Analysis 1: Comparison: Placebo; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in FS at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.3748, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = 0.95, 95% CI 2-sided [-1.204 to 3.102]

10. Secondary Outcome: Post-baseline Changes Compared to Placebo (at 1-, 2-, and 3-hours Post Infusion Initiation [ie, at the End of 5, 15 and 30 ng/kg/Min Infusions]) in Stroke Volume (SV)
Description: The primary analysis of this study focused on the differences between the treatment groups in terms of Least Squares (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from Baseline in Stroke Volume (SV) at the end of the 30 ng/kg/min infusion as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL/beat
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 16 | 44
mL/beat
  1 hour infusion (5 ng/kg/min) | -1.34 (6.51) [-4.198 to 18.359] | 5.75 (4.84)
  2 hour infusion (15 ng/kg/min) | -4.33 (6.23) [-2.016 to 19.575] | 4.45 (4.63)
  3 hour infusion (30 ng/kg/min) | -0.62 (6.7) [2.557 to 25.771] | 13.54 (4.98)
Statistical Analysis 1: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in SV at the end of the 5 ng/kg/min dose; Test type: Superiority or Other; p = 0.2123, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = 7.08, 95% CI 2-sided [-4.198 to 18.359]
Statistical Analysis 2: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in SV at the end of the 15 ng/kg/min dose; Test type: Superiority or Other; p = 0.1083, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = 8.78, 95% CI 2-sided [-2.016 to 19.575]
Statistical Analysis 3: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in SV at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.0180, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = 14.16, 95% CI 2-sided [2.557 to 25.771]

11. Secondary Outcome: Post-baseline Changes Compared to Placebo (at 1-, 2-, and 3-hours Post Infusion Initiation [ie, at the End of 5, 15 and 30 ng/kg/Min Infusions]) in Pulmonary Arterial Systolic Pressure (PASP)
Description: The primary analysis of this study focused on the differences between the treatment groups in terms of Least Squares (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from Baseline in Pulmonary Arterial Systolic Pressure (PASP) at the end of 5, 15 and 30 ng/kg/min Infusions as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 16 | 46
mmHg
  1 hour infusion (5 ng/kg/min) | 2.69 (2.10) [-5.308 to 2.554] | 1.32 (1.55)
  2 hour infusion (15 ng/kg/min) | 0.51 (2.45) [-5.567 to 3.594] | -0.48 (1.80)
  3 hour infusion (30 ng/kg/min) | -0.79 (2.74) [-4.107 to 6.148] | 0.24 (2.02)
Statistical Analysis 1: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in PASP at the end of the 5 ng/kg/min dose; Test type: Superiority or Other; p = 0.4841, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-5.308 to 2.554]
Statistical Analysis 2: Comparison: Placebo vs JNJ-39588146; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; p = 0.6665, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-5.567 to 3.594]
Statistical Analysis 3: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in PASP at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.6904, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = 1.02, 95% CI 2-sided [-4.107 to 6.148]

12. Secondary Outcome: Post-baseline Changes Compared to Placebo (at 1-, 2-, and 3-hours Post Infusion Initiation [ie, at the End of 5, 15 and 30 ng/kg/Min Infusions]) in Pulmonary Arterial Diastolic Pressure (PADP)
Description: The primary analysis of this study focused on the differences between the treatment groups in terms of Least Square (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from Baseline in Pulmonary Arterial Diastolic Pressure (PADP) at the end of 5, 15 and 30 ng/kg/min Infusions as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 16 | 46
mmHg
  1 hour infusion (5 ng/kg/min) | -0.99 (1.57) [-2.197 to 3.558] | -0.29 (1.12)
  2 hour infusion (15 ng/kg/min) | -0.83 (1.91) [-3.851 to 3.153] | -1.17 (1.36)
  3 hour infusion (30 ng/kg/min) | -0.72 (1.85) [-4.138 to 2.669] | -1.46 (1.32)
Statistical Analysis 1: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in PADP at the end of the 5 ng/kg/min dose; Test type: Superiority or Other; p = 0.6304, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = 0.70, 95% CI 2-sided [-2.197 to 3.588]
Statistical Analysis 2: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in PADP at the end of the 15 ng/kg/min dose; Test type: Superiority or Other; p = 0.8420, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-3.851 to 3.153]
Statistical Analysis 3: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in PADP at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.6658, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-4.138 to 2.669]

13. Secondary Outcome: Post-baseline Changes Compared to Placebo (at 1-, 2-, and 3-hours Post Infusion Initiation [ie, at the End of 5, 15 and 30 ng/kg/Min Infusions]) in Calculated Systemic Vascular Resistance (SVR)
Description: The primary analysis of this study focused on the differences between the treatment groups in terms of Least Squares (LS) mean change from Baseline at each time point; thus, the results provided below consist of the JNJ-39588146 minus placebo differences in LS means (and associated confidence intervals) for change from Baseline in Calculated Systemic Vascular Resistance (SVR) at the end of 5, 15 and 30 ng/kg/min Infusions as well as treatment group LS means and Standard Errors.
Time Frame: Baseline up through 3 hours post infusion initiation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: dyn.s.cm-5
Arm/Group | Placebo | JNJ-39588146
Number analyzed (Participants) | 14 | 45
dyn.s.cm-5
  1 hour infusion (5 ng/kg/min) | 67.41 (147.97) [-529.875 to 1.147] | -196.95 (105.33)
  2 hour infusion (15 ng/kg/min) | 321.97 (116.73) [-592.781 to -173.867] | -61.36 (83.09)
  3 hour infusion (30 ng/kg/min) | 281.79 (131.69) [-764.070 to -291.478] | -245.98 (93.74)
Statistical Analysis 1: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in SVR at the end of the 5 ng/kg/min dose; Test type: Superiority or Other; p = 0.0510, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -264.36, 95% CI 2-sided [-529.875 to 1.147]
Statistical Analysis 2: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in SVR at the end of the 15 ng/kg/min dose; Test type: Superiority or Other; p = 0.0006, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -383.32, 95% CI 2-sided [-592.781 to -173.867]
Statistical Analysis 3: Comparison: Placebo vs JNJ-39588146; 95% confidence intervals and p values represent the placebo-subtracted LS mean change from baseline in SVR at the end of the 30 ng/kg/min dose; Test type: Superiority or Other; p = 0.0001, ANCOVA — two-sided p-value and two-sided alpha=0.05; Mean Difference (Final Values) = -527.77, 95% CI 2-sided [-764.070 to -291.478]

ADVERSE EVENTS:
Time Frame: The number of patients with serious adverse events (SAEs) and other adverse events reported from the time of the first dose of study drug through the last examination/follow-up visit or 4 weeks after dosing are provided in the table below.
Description: One SAE of Cardiac Failure in the JNJ-39588146 group classified as non-treatment emergent was verified as "treatment-emergent" after database lock. Thus, 3(7%) patients in the JNJ-39588146 group experienced a treatment-emergent SAE of Cardiac Failure and the total number of patients with treatment-emergent SAEs in the JNJ-39588146 group was 6(13%).
Arm/Group | Placebo | JNJ-39588146
Serious Adverse Events (participants affected / at risk) | 3/16 | 5/46
Other Adverse Events (participants affected / at risk) | 8/16 | 11/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | JNJ-39588146 (N=46)
Cardiac Failure (Cardiac disorders) | 1 | 2
Cardiac Arrest (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Device Malfunction (General disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | JNJ-39588146 (N=46)
Ventricular Tachycardia (Cardiac disorders) | 1 | 2
Cardiac Failure (Cardiac disorders) | 1 | 1
Ventricular Arrhythmia (Cardiac disorders) | 1 | 1
Ventricular Extrasystoles (Cardiac disorders) | 2 | 0
Feeling Hot (General disorders) | 0 | 3
Pyrexia (General disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 2
Tooth Disorder (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Flushing (Vascular disorders) | 2 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Data from the extended infusion sub-study were exploratory; therefore, results for outcome measures from the sub-study are not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator wishes to publish information from the study, a copy of the manuscript must be provided to the Sponsor for review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the Sponsor in writing, the Investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.